CLINICAL TRIAL: NCT00629863
Title: Cancer of the Oesophagus or Gastricus: New Assessment of the Technology of Endosonography COGNATE
Brief Title: Endoscopic Ultrasound in Diagnosing Cancer in Patients With Localized Stomach Cancer or Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Wales Organisation for Randomised Trials in Health (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: NWORTH-COGNATE; CDR0000584174 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN01444215; NWORTH-04/MRE10/10
Record Dates: First submitted 2008-03-05; First posted 2008-03-06 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-01

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Cisplatin; Fluorouracil; Neoadjuvant Therapy; High-Energy Shock Waves; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Other: questionnaire administration
Procedure: diagnostic endoscopic procedure
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery
Procedure: therapeutic endoscopic surgery
Procedure: ultrasound imaging
Radiation: radiation therapy
Radiation: radioisotope therapy

SUMMARY:
RATIONALE: Diagnostic procedures, such as endoscopic ultrasound, may help doctors learn the extent of stomach cancer or esophageal cancer.

PURPOSE: This randomized clinical trial is studying how well endoscopic ultrasound works in diagnosing cancer in patients with localized stomach cancer or esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the additional effect of endoscopic ultrasound (EUS) staging compared with a standard staging algorithm on the selection of treatment in patients with gastric or esophageal cancer (GOC), including the numbers of patients treated surgically, with multimodality therapy, or with non-surgical means.
* To estimate the effect of EUS staging on the outcome of care of these patients.
* To assess the cost-effectiveness of EUS by comparing improvements in patient outcomes with the additional costs of the procedure.
* To estimate the proportion of patients with GOC who will benefit from EUS and therefore to determine the need for EUS facilities within a population.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor location (gastric vs esophageal vs gastroesophageal junction) and participating center.

All patients undergo standard staging methods. Patients with localized tumors are randomized to undergo either endoscopic ultrasound (EUS) or no further staging. Both groups receive treatment as follows, depending on the type of tumor:

* Mucosal tumors: Patients undergo endoscopic mucosal resection and argon-beam ablation of the surrounding mucosa.
* Resectable tumors: Patients undergo surgery and neoadjuvant chemotherapy comprising cisplatin and fluorouracil.
* Advanced localized disease without the possibility of complete resection: Patients receive chemoradiotherapy or chemotherapy alone depending upon the site. Patients with gastric cancer may undergo palliative surgery.

Quality of life is assessed at 1, 3, 6, 12, 18, and 24 months using questionnaires, including the EuroQol EQ-5D, the EORTC core module QLQ-C30, the EORTC esophageal module QLQ-OES24, and the EORTC gastric module QLQ-STO22.

After completion of study treatment, patients are followed every 3 months for a minimum of 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of gastric or esophageal cancer

  * Localized disease
  * No metastatic disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* American Society of Anesthesiologists grade 1 (no physiological disturbance) or 2 (minor well-compensated physiological impairment)
* Must be fit for surgery and chemotherapy

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Overall survival at 12 months of patients last randomized and at 48 months of patients first randomized

SECONDARY OUTCOMES:
Complete resection rate
Quality of survival in the different treatments selected on the basis of staging at 1, 3, 6, 12, 18, and 24 months by EuroQol EQ-5D, EORTC core module QLQ-C30, EORTC esophageal module QLQ-OES24, and EORTC gastric module QLQ-STO22
Health resource utilization, including the selection of treatments and subsequent use of health service resources

CONTACTS AND LOCATIONS:
Overall Officials: Ken Park, MD, Study Chair — North Wales Organisation for Randomised Trials in Health
Locations (9):
- United Kingdom (9):
  - Royal Blackburn Hospital, Blackburn, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Leicester Royal Infirmary, Leicester, England
  - North Tyneside Hospital, North Shields, England
  - Southampton General Hospital, Southampton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - North Wales Organisation for Randomised Trials in Health, Bangor, Wales